CLINICAL TRIAL: NCT06579170
Title: Burden of Recreational Water Illness Due to Exposure to Cyanobacteria and Their Toxins in Freshwater Beaches in Canada: a Prospective Cohort Study
Brief Title: Burden of Recreational Water Illness Due to Exposure to Cyanobacteria and Their Toxins in Freshwater Beaches in Canada
Status: Active, not recruiting | Type: Observational
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Ontario Ministry of the Environment, Conservation and Parks (Unknown); Manitoba Environment and Climate Change (Unknown); Windsor-Essex County Health Unit (Unknown); Canadian Veterinary Medical Association (Unknown); Health Canada (Other Government)
Responsible Party: Principal Investigator, Ian Young, Associate Professor, Toronto Metropolitan University
Other Study IDs: 2324-HQ-000024
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Gastroenteritis; Gastrointestinal Diseases; Eye Infections; Skin Infections; Respiratory Tract Infections; Blue Green Algae Poisoning
Keywords: Cohort study; Harmful algal blooms; Recreational water contact; Cyanobacteria; One Health
MeSH Terms: conditions — Gastroenteritis; Gastrointestinal Diseases; Eye Infections; Cellulitis; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Recreational water users: Recreational water users of any age and their pet dogs present at the beaches and waterfronts in this study during recruitment days.
  Interventions: Behavioral: Cyanobacteria exposure during water contact

INTERVENTIONS:
Behavioral: Cyanobacteria exposure during water contact — Cyanobacteria levels in beach water among participants who report water contact in the beach survey

SUMMARY:
Swimming and other recreational water activities at public beaches are increasingly popular leisure activities among Canadians. However, harmful algal blooms caused by blue-green algae (i.e., cyanobacteria) have also been increasing reported at Canadian public beaches in recent years. These algal blooms can cause various acute illnesses among recreational water users through ingestion, inhalation of aerosols, or skin contact with contaminated water. In addition, blue-green algae blooms and their toxins can cause illnesses in pets and wildlife. Currently, baseline data are lacking on the risk of recreational water illness from exposure to blue-green algae blooms in Canada. This study will identify the burden of recreational water illness among recreational water users at four targeted beach sites in Ontario, Manitoba and Nova Scotia, over a two-year period. A prospective cohort study design will be used. The investigators will determine the risk of acquiring acute illness outcomes in recreational water users, as well as their pet dogs, that engage in different levels of water contact at beaches at risk of blue-green algae blooms. The investigators will examine differences in illness risks by gender, age, and location. Relationships between cyanobacterial cell counts, toxin levels, and environmental conditions with the risk of acute illness among participants will be determined. Overall, results will provide important data on the risk of recreational water illness from exposure to blue-green algae and their toxins in Canadian beach settings.

DETAILED DESCRIPTION:
This study will investigate the incidence of recreational water illness due to exposure to cyanobacterial blooms and their toxins in four targeted and popular freshwater beaches in Ontario, Manitoba, and Nova Scotia, Canada. A prospective cohort design and One Health approach will be used. On-site recruitment of recreational water users will be conducted at two beaches per year during the summers of 2024 and 2025. The population of interest includes recreational water users of any age and their pet dogs. After enrollment, an in-person survey will determine beach exposures and confounding factors, and a three-day follow-up survey will ascertain any acute illness outcomes experienced by participants or their dogs. The target sample size is 2500 recreational water users. Water samples will be taken each recruitment day and analyzed for cyanobacterial indicators (pigments), cell counts, and toxin levels. Regression analysis will be conducted to estimate the association with water contact, cyanobacterial levels, and risks of different acute illness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent
* ability to complete the surveys in English or French
* must not have participated in the study in the past 21 days

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recreational water users of any age, and any pet dogs also present at the beaches/waterfront areas, during the study recruitment days.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of gastrointestinal illness among participants | Within 3 days of beach visit
  Gastrointestinal illness is defined as one or more of: (a) diarrhea (≥3 loose stools in 24 hrs); (b) vomiting; (c) nausea with stomach cramps; or (d) nausea or stomach cramps that interfere with regular daily activities (e.g., missed work or school)

SECONDARY OUTCOMES:
Incidence of respiratory illness among participants | Within 3 days of beach visit
  Defined as: sore throat, runny or congested nose, difficulty breathing, or cough
Incidence of eye infections among participants | Within 3 days of beach visit
  Defined as: eye infection or irritation
Incidence of skin infections among participants | Within 3 days of beach visit
  Defined as: rash or itchy skin
Incidence of generalized symptoms among participants | Within 3 days of beach visit
  Defined as: headache, fever, fatigue, dizziness, loss of appetite, chills, muscle pain, or general pain

OTHER OUTCOMES:
Incidence of illness severity measures among participants | Within 3 days of beach visit
  Medical consultations, hospital visits, medication use, and hospitalization

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Grand Beach, Winnipeg, Manitoba
  - Shubenacadie Canal, Halifax, Nova Scotia
  - Kinsmen beach, Port Perry, Ontario
  - Colchester Beach, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: Yes
An anonymized dataset will be shared publicly after results are published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Study protocol is already published. Code and dataset will be shared after study publication of results.
URL: https://doi.org/10.1136/bmjopen-2024-085406

REFERENCES:
- [Background] Young I, Sanchez JJ, Sekerciouglu F, Desta BN, Holeton C, Lyng D, Peczulis V, Renwick S, Brooks T, Tustin J. Burden of recreational water illness due to exposure to cyanobacteria and their toxins in freshwater beaches in Canada: protocol of a prospective cohort study. BMJ Open. 2024 Jun 12;14(6):e085406. doi: 10.1136/bmjopen-2024-085406. PMID 38866574